CLINICAL TRIAL: NCT06393166
Title: An Open-label, Single-arm, Multicenter, Phase II Clinical Study of the Efficacy and Safety of Sequential AG and mFOLFOX Combined With Serplulimab Injection and Bevacizumab Injection in Patients With Untreated Advanced Pancreatic Cancer
Brief Title: Sequential AG and mFOLFOX Combined With Serplulimab Injection and Bevacizumab Injection in Untreated Advanced Pancreatic Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Principal Investigator, Ying Jieer, Chief physician, Zhejiang Cancer Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-2023-384
Record Dates: First submitted 2024-04-28; First posted 2024-05-01 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2024-04

CONDITIONS: Non-Resectable Pancreas Carcinoma
MeSH Terms: interventions — Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sequential AG and mFOLFOX in Combination With Serplulimab Injection and Bevacizumab Injection (Experimental): Nab-paclitaxel:125 mg/m2, ivgtt, D1, 8 and 15,every 6 weeks for a treatment cycle Gemcitabine hydrochloride: 1g/m2, ivgtt, D1, 8 and 15,every 6 weeks for a treatment cycle 5-FU: 2400 mg/m2 ,ivgtt over 46h, D29-30, every 6 weeks for a treatment cycle Oxaliplatin: 85 mg/m2 ,ivgtt, D29, every 6 weeks for a treatment cycle LV: 400 mg/m2 ,ivgtt over 2h, D29, every 6 weeks for a treatment cycle Serplulimab Injection: 3mg/kg,ivgtt,D1, every 2 weeks for a treatment cycle. Bevacizumab Injection: 5mg/kg,ivgtt,D1, every 2 weeks for a treatment cycle.
  Interventions: Drug: Sequential AG and mFOLFOX in Combination With Serplulimab Injection and Bevacizumab Injection

INTERVENTIONS:
Drug: Sequential AG and mFOLFOX in Combination With Serplulimab Injection and Bevacizumab Injection — Nab-paclitaxel:125 mg/m2, ivgtt, D1, 8 and 15,every 6 weeks for a treatment cycle Gemcitabine hydrochloride: 1g/m2, ivgtt, D1, 8 and 15,every 6 weeks for a treatment cycle 5-FU: 2400 mg/m2 ,ivgtt over 46h, D29-30, every 6 weeks for a treatment cycle Oxaliplatin: 85 mg/m2 ,ivgtt, D29, every 6 weeks for a treatment cycle LV: 400 mg/m2 ,ivgtt over 2h, D29, every 6 weeks for a treatment cycle Serplulimab Injection: 3mg/kg,ivgtt,D1, every 2 weeks for a treatment cycle. Bevacizumab Injection: 5mg/kg,ivgtt,D1, every 2 weeks for a treatment cycle.

SUMMARY:
It is a single arm, open-label, multicenter, phase II cinical trial to evaluate the efficacy and safety of the Sequential AG and mFOLFOX in Combination With Serplulimab Injection and Bevacizumab Injection in first-line treatment of patients with Advanced or Metastatic Pancreatic Cancer.

DETAILED DESCRIPTION:
It is a single arm, open-label, multicenter, phase II cinical trial to evaluate the efficacy and safety of the Sequential AG and mFOLFOX in Combination With Serplulimab Injection and Bevacizumab Injection in first-line treatment of patients with Advanced or Metastatic Pancreatic Cancer. A Simon two-stage study design was utilized. Treatment will continue until disease progression or toxicity is intolerable. The plan is to enroll 37 subjects in multiple hospitals in china.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily agree to participate in the study and sign the informed consent;
2. ≥18 years of age and ≤75 years of age on the day of signing the informed consent form, regardless of gender;
3. Pancreatic ductal adenocarcinoma confirmed by pathologic histology or cytology;
4. No prior systemic therapy for unresectable locally advanced or metastatic pancreatic cancer;
5. Measurable lesions at baseline according to RECIST 1.1 criteria; if the subject has only 1 measurable lesion at baseline, the area of the lesion must not have received radiotherapy in the past or there must be evidence of significant progression of the lesion after completion of radiotherapy treatment;
6. the ECOG physical status score was 0 or 1 and the Expected survival ≥12 weeks;
7. No serious organic diseases of the heart, lungs, brain and other organs;
8. Adequate organ function

   1. Bone Marrow Function: (no transfusion within 14 days prior to screening, no use of granulocyte colony stimulating factor [G-CSF], no use of drug correction) : i. Hemoglobin ≥90g/L; ii. Leukocytes ≥ 4.0 x 109/L, Neutrophils ≥1.5×109/L; iii. Platelet ≥80×109/L;
   2. Coagulation function: PT or APTT ≤ 1.5 x ULN in subjects not receiving anticoagulation; if subjects are receiving anticoagulation, as long as the PT is within the range of the anticoagulant drug formulation;
   3. liver function: (no albumin infusion within 14 days prior to screening): Serum total bilirubin ≤ 1.5 x ULN (with biliary obstruction, allowing enrollment of subjects undergoing biliary drainage or in the midst of stenting therapy who have a total bilirubin ≤ 2.5 x ULN). In subjects without liver metastasis, Aspartate aminotransferase (AST), alanine aminotransferase (ALT)≤2.5×ULN; In subjects with liver metastasis, ALT and AST≤5×ULN, but without elevated bilirubin;
   4. Renal function: serum creatinine ≤1.5 x ULN, creatinine clearance (CCr) ≥50 mL/min, urinary protein <2+ (if urinary protein ≥2+, 24-hour (h) urinary protein quantification can be carried out, and 24h urinary protein quantification <1.0 g can be enrolled)
   5. Heart function: New York College of Cardiology (NYHA) rating < 3; Left ventricular ejection fraction ≥50%;
9. Male or female patients of childbearing potential will voluntarily use an effective method of contraception, such as a double-barrier contraceptive method, condoms, oral or injectable contraceptives, and an intrauterine device (IUD), for the duration of the study and up to 6 months after the last study dose. All female patients will be considered of childbearing potential unless the female patient is naturally menopausal, artificially menopausal or sterilized;
10. Subject's ability and willingness to comply with visits, treatment plans, laboratory tests, and other study-related processes as specified in the study protocol.

Exclusion Criteria:

1. subjects with clear brain metastases on imaging or with meningeal metastases;
2. untreated spinal compression fractures not treated by surgery and/or radiotherapy; treated spinal compression fractures require disease stabilization for at least 2 weeks prior to enrollment;
3. high risk of gastrointestinal or abdominal bleeding as evaluated by the Investigator;
4. uncontrolled cancer pain; narcotic analgesics not at a stable dose at enrollment;
5. previous treatment with vascular endothelial growth factor (VEGFR) inhibitors or previous treatment with immune checkpoint inhibitors;
6. antitumor treatment with chemotherapy, small molecule inhibitors, immunotherapy (e.g., interleukin, interferon, or thymosin) within 28 days prior to enrollment in this study, and herbal medicine with antitumor indications within 14 days prior to dosing;
7. major surgical procedures [such as transabdominal, transthoracic and other major surgeries; excluding diagnostic puncture such as ultrasonic endoscopy-guided pancreatic fine-needle aspiration biopsy (EUS-FNB), percutaneous hepatic perforation biopsy, peripheral venous catheterization, and biliary stent implantation] or invasive treatments or operations with incomplete healing of the surgical incision, local anti-tumor treatment such as hepatic artery interventional embolization, hepatic metastasis cryo-ablation, radiofrequency ablation and other local anti-tumor treatments. radiofrequency ablation and other local antitumor therapy;
8. have received radical radiotherapy within 3 months prior to study entry; palliative radiotherapy 2 weeks prior to dosing is permitted, and the dose of radiotherapy meets local standards of care for palliative care;
9. required systemic corticosteroid (>10 mg/day prednisone or equivalent of other corticosteroid for ≥7 consecutive days) or immunosuppressive therapy within 14 days prior to enrollment in this study; with the exception of inhaled or locally applied hormones, or physiologic replacement doses of hormone therapy due to adrenal insufficiency; short-term (≤7 days) corticosteroids are allowed for prophylaxis (e.g., contrast allergy) or treatment of Non-autoimmune conditions (eg, delayed hypersensitivity reactions caused by exposure to allergens) ;
10. subjects with uncorrectable albumin decline (serum albumin <3.0 g/dL) 14 days prior to enrollment in this study; and
11. a 10% or greater weight loss in comparison to the weight loss at the time of ICF signing within 72 hours prior to enrollment in this study; and
12. within 72 hours prior to study entry, the subject's ECOG physical status score increases by ≥1 point compared to the ICF score; 13. within 28 hours prior to study entry, the subject's ECOG physical status score increases by ≥1 point compared to the ICF score; and
13. has received a live vaccine (including live attenuated vaccine) within 28 days prior to enrollment in this study;
14. previous or current interstitial pneumonia/pneumatosis, unless determined by the investigator to be inactive and not requiring hormonal therapy; and
15. pre-existing or current autoimmune disease, including but not limited to Crohn's disease, ulcerative colitis, systemic lupus erythematosus, tuberculosis, Wegener's syndrome (granulomatous disease with polyangiitis), Graves' disease, rheumatoid arthritis, hypopituitarism, uveitis, autoimmune hepatitis, systemic sclerosis ( Scleroderma, etc.), Hashimoto's thyroiditis, autoimmune vasculitis, autoimmune neuropathy (Guillain-Barre syndrome). The following conditions are excluded: type I diabetes mellitus, hypothyroidism stabilized by hormone replacement therapy (including hypothyroidism caused by autoimmune thyroid disease), psoriasis or vitiligo that does not require systemic therapy;
16. a combination of other malignancies within the last 5 years, except cured squamous skin cancer, basal cell carcinoma, non-basal invasive bladder cancer, and prostate/cervical/breast cancer in situ;
17. hepatic metastases comprising more than 50% of the total liver volume;
18. uncontrolled comorbidities, including but not limited to the following

    1. Active HBV or HCV infection; (Note: HBV DNA and/or HCV RNA testing is required for subjects who are HBsAg positive and/or HCV antibody positive at Screening. Subjects who are negative for HBV DNA ≤500 IU/mL (or ≤2000 copies/mL) and/or HCV RNA are eligible for enrollment; HBsAg-positive subjects are required to have their HBV DNA monitored during the course of treatment);
    2. Known history of HIV infection or AIDS;
    3. Active syphilis;
    4. Active tuberculosis;
    5. Active or uncontrolled serious infection (≥ CTCAE grade 2 infection);
    6. Medication-uncontrolled hypertension (defined as systolic blood pressure ≥140 mmHg and/or diastolic blood pressure ≥90 mmHg;), symptomatic cardiac insufficiency (NYHA II-IV), unstable angina pectoris or myocardial infarction within 6 months, or the presence of a prolonged QTc or risk of torsades de pointes (baseline QTc>470 msec (women)/450 msec (men) < Fridericia method correction>, hypokalemia, long QT syndrome, atrial fibrillation with heart rate >100 bpm at rest or severe cardiac valvular disease, history of medically significant arrhythmias);
19. unrecovered toxicity from prior antitumor therapy to CTCAE ≤ Grade 1 (NCI-CTCAE v5.0), except for baldness (any grade allowed) and peripheral neuropathy (recovery to ≤ Grade 2 required);
20. history of prior allogeneic bone marrow or organ transplantation;
21. prior history of allergic reaction, hypersensitivity reaction, intolerance to investigational drugs or similar medications; prior significant allergy to drugs or foods or other substances (e.g., severe allergic reaction, immune-mediated hepatotoxicity, immune-mediated thrombocytopenia, or anemia)
22. pregnant and/or lactating women;
23. other conditions that, in the opinion of the investigator, would affect the safety of or adherence to treatment with the study medication, including alcoholism, drug abuse, other serious illnesses (including psychiatric illnesses) that require comorbid treatment, the presence of serious laboratory test abnormalities, moderate to large amounts of plasmapheresis such as pleural fluid, pericardial effusion, ascites, and other concomitant familial or social factors, which would affect the safety of the patient;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective response rate(ORR) | [ up to 12 months]
  The number of cases in which tumor size is reduced to PR or CR / the total number of evaluable cases (%)

SECONDARY OUTCOMES:
Progression-free survival (PFS) | [ up to 12 months]
  Refers to the date from the date of admission to the date of the first progression of disease or death of any cause, using Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1).
Overall survival (OS) | [ up to 36 months]
  The time interval between the start date of study drug and the date of death (any cause)
Disease control rate (DCR) | [ up to 12 months]
  Percentage of confirmed cases including complete remission (CR), partial remission (PR) and disease stability (SD) among patients with evaluable efficacy
Incidence of Treatment-Emergent 3/4 Adverse Events | [up to 12 months after enrollment or study close]
  Number and percentage of participants with Adverse Events (any Grade and Grade 3/4)

OTHER OUTCOMES:
Blood or tissue biomarkers | [up to 12 months after enrollment or study close]
  Detection of PD-L1 Expression by Immunohistochemistry; Gene Level Changes in Tissues by Single Cell Sequencing; Peripheral Blood Lymphocyte Subpopulations by Flow Cytometry

CONTACTS AND LOCATIONS:
Overall Officials: Jieer Ying, Principal Investigator — Zhejiang Cancer Hospital
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No